CLINICAL TRIAL: NCT06905067
Title: Assessment of Oral Health in Minors Incarcerated at Fleury Merogis: Retrospective Observational Study
Acronym: DENTMIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0007
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: DMFT Index, ICDAS Score, Dental Plaque Index, Communication, Prevention, Dentist, Orthodontist
Keywords: dental caries; DMF index; oral health; oral hygiene; humans; adolescent; jails; prisoners; young adult; male; prevalence; france; epidemiology; retrospective studies; observational studies as topic
MeSH Terms: conditions — Communication; Dental Caries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Minors incarcerated in fleury-Merogis prison: male minors incarcerated in fleury merogis prison for a period between June and December 2024.
  Interventions: Other: questionnaire and dental clinical examination

INTERVENTIONS:
Other: questionnaire and dental clinical examination — Assessment of the DMFT index

SUMMARY:
The goal of this study is to assess the oral health of males juveniles incarcerated at Fleury-Mérogis over a given period.

The goal is also to understand the needs of these patients and improve their care in prison while raising awareness about oral health to achieve lasting results.

Hypothesis: Incarcerated juveniles often grew up in precarious conditions. Is their DMFT (decayed, missing, filled permanent teeth) index higher than the "standard" juvenile population? Public interest: Understanding the needs of these juvenile patients, public health data.

By comparing our results to those of the "standard" population (non-incarcerated minors) through a literature review regarding the DMFT index in these patients, we will determine whether incarcerated juvenile patients represent a population at risk of developing oral pathologies. Oral disease prevention for these patients to raise awareness of the importance of oral hygiene and follow-up dental appointments outside of the prison system. The earlier these patients are educated, the greater the chance they will develop better habits throughout their lives.

DETAILED DESCRIPTION:
This is a retrospective observational study in which we will collect data from the first dental consultation between June 2024 and December 2024.

The primary objective is to assess the oral health of minors incarcerated at Fleury-Mérogis using the primary outcome measure, the DMFT index.

77 male minors are included in the study. Data will be collected retrospectively by the research team from their medical records.

The data will be collected by the research team in a pseudo-anonymized form in an electronic CRF (case report form) and then analyzed by the biostatistician at the Clinical Research Unit of the Centre Hospitalier Sud Francilien.

ELIGIBILITY:
Inclusion Criteria:

* Male minor patients incarcerated at the Fleury-Mérogis Prison between June 2024 and December 2024
* Patients who have had a dental check-up

Exclusion Criteria:

- Patients and/or those with parental authority who have been informed and have objected to the use of their data.- Female patients and/or those with parental authority over the newborn who have objected to the use of their data.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: male minors incarcerated in Fleury-Mérogis over the study period (between June 2024 and December 2024)
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Decayed missing filled permanent teeth index (DMFT | at day 0
  Number of decayed, missing and filled permanent teeth

SECONDARY OUTCOMES:
Frequency of brushing and presence of absence of snacking | at day 0
  Assess oral hygiene and dietary habits
NRS scale | at day 0
  NRS (numeric rating scale) : A score of 0 means no pain, and 10 means the worst pain you have ever felt.
Presence of oral pathology defined by a DMFT index > 0 | at day 0
  Assess oral pathologies in incarcerated minors

CONTACTS AND LOCATIONS:
Overall Officials: Dominique ORPHELIN, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No